CLINICAL TRIAL: NCT06950866
Title: Home-Based Executive Function Training Intervention For Attention-Deficit/ Hyperactivity Disorder-prone Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan Mental Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2024.0710.15
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: Attention Deficit Hyperactivity Disorder (ADHD); Executive function training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Home-based executive function training therapy
- Waitlist group (Other)
  Interventions: Behavioral: Home-based executive function training therapy

INTERVENTIONS:
Behavioral: Home-based executive function training therapy — Parents receive a 2-week, 20-session online child executive function training program, delivered by a systematically trained and supervised therapist.
  Arms: Intervention group
Behavioral: Home-based executive function training therapy — After the postintervention data collection, parents in the waitlist group receive a 2-week, 20-session online child executive function training program, delivered by a systematically trained and supervised therapist.
  Arms: Waitlist group

SUMMARY:
This study aims to investigate the effectiveness of a home-based executive function training Intervention on children's ADHD symptoms, executive function and parents' parenting stress.

ELIGIBILITY:
Inclusion Criteria:

* 1.SNAP-IV scale, inattention or hyperactivity-impulsivity scale score > 1.2
* 2.Parents who could understand or lacking of access to computers and the Internet
* 3.Parents can commit to ensuring full participation and complete the training and test evaluations in full compliance with the researcher's requirements
* 4.Children and their parents consent to the study

Exclusion Criteria:

* 1.Children or parents with severe organic encephalopathy and other severe mental disorders
* 2.Parents or children are receiving ADHD-related behavioral treatment
* 3.Parents or children who dropped out before the study started or in the middle of the study

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
1.Chinese version of Swan-son Nolan and Pelham, Version IV Scale-parent form (SNAP-IV) | Baseline, 1 month after intervention, 2 months after intervention
  This questionnaire is used to evaluate the children's ADHD symptoms.
2.Behavior Rating Inventory of Executive Function (BRIEF) | Baseline, 1 month after intervention, 2 months after intervention
  This questionnaire is used to evaluate the children's executive function.
3.Parenting Stress Index-Short Form (PSI-SF) | Baseline, 1 month after intervention, 2 months after intervention
  This questionnaire is used to evaluate the parents' parenting stress.

SECONDARY OUTCOMES:
4.Client Satisfaction Questionnaire (CSQ) | Baseline, 1 month after intervention, 2 months after intervention
  This questionnaire is used to evaluate the parents' satisfaction with the intervention.